CLINICAL TRIAL: NCT01776918
Title: Energy Requirements in Metabolic and Mitochondrial Disease
Brief Title: Energy Requirements in Mitochondrial Disease
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Rare Disease Foundation, Vancouver, Canada (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Other Study IDs: H11-02094
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Mitochondrial Disease; Chronic Metabolic Disorder
Keywords: POLG1 Mutation; Phenylketonuria
MeSH Terms: conditions — Mitochondrial Diseases; Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metabolic Disease- Phenylketonuria
- Mitochondrial disorder

SUMMARY:
Metabolic diseases and mitochondrial disorders are caused by genetic mutation which lead to disruptions in energy producing pathways in our body. Enough energy or calories must be given in the diet to ensure normal growth and development. Currently, energy needs for patients with metabolic and mitochondrial diseases are not measured, but is estimated using a mathematical equation based on healthy children. This may lead to under feeding or overfeeding of calories, and has negative nutritional implications.

The clinical standard for measuring energy needs is the use of indirect calorimeter.The indirect calorimeter takes individualized measurements for each patient and therefore will enable dietitians and clinicians to provide sufficient calories in the diet to better manage the disease and promote normal growth and development.

We believe daily energy requirements will vary within metabolic diseases (Phenylketonuria) and mitochondrial disorders (mitochondrial fatty acid oxidation defect, POLG1 mutation etc.).

The objective of this preliminary study is to measure resting energy expenditure in children living with metabolic and mitochondrial conditions and data obtained will be used to generate future hypothesis and will form a basis for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Children(1-18y) who are diagnosed with either Phenylketonuria (PKU) or a mitochondrial disorder

Exclusion Criteria:

* Children, less than 1y old, who are diagnosed with PKU or a mitochondrial disorder, as it is difficult to perform indirect calorimeter on them.
* Children(1-18y) who are not diagnosed with PKU or a mitochondrial disorder
* Children(1-18y) who are diagnosed with either PKU or a mitochondrial disorder, but are currently experiencing illness such as fever, cold, vomiting or diarrhea

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (1-18y) diagnosed with either phenylketonuria or a mitochondrial disorder
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | 1 hour
  Resting Energy Expenditure will be measured by carbon dioxide production and oxygen consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — Child & Family Research Institute/University of British Columbia; Sylvia Stockler-Ipsiroglu, Study Chair — University of British Columbia/Faculty of Pediatrics; Ramona Meni Salvarinova Zivkovic, Study Chair — University of Bristish Columbia/Faculty of Pediatrics; Howard Parsons, Study Chair — University of British Columbia/Faculty of Pediatrics
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada